CLINICAL TRIAL: NCT01468857
Title: A Pilot Study to Examine Physiological and Clinical Markers of Chronic Stress in Caregivers of Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients
Brief Title: Physical and Emotional Health of Caregivers for People Who Have Had Stem Cell Transplants
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110265; 11-CC-0265
Record Dates: First submitted 2011-10-06; First posted 2011-11-10 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-09-28

CONDITIONS: Stress; Family Caregivers
Keywords: Clinical Stress Markers; Chronic Stress; Allogeneic Hematopoietic Stem Cell Transplant; HSCT Caregivers; Cancer Caregivers; Stress; Family Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Stem cell transplants are a complex treatment that can have serious side effects. Having a caregiver to help with the recovery is critical. Serving in this role, however, can cause high stress levels and negative health effects. Researchers want to better understand the health effects of caring for a family member or friend after a stem cell transplant. Understanding these effects can help develop programs that support caregivers coping with the demands of post-transplant care.

Objectives:

- To study the physical and emotional health of caregivers for a family member or friend who has had a stem cell transplant.

Eligibility:

* Individuals at least 18 years of age who are planning to be a caregiver for a person having a stem cell transplant.
* Healthy non-caregiver volunteers for comparison studies.

Design:

* A caregiver will be caring for a transplant recipient just before transplant admission and up through 6 weeks after hospital discharge. The caregiver will usually live with or spend at least 6 hours each day with the recipient.
* All participants will have three study visits. The first visit will happen before the transplant. The second and third visits will happen at the recipient s discharge, and 6 weeks after discharge. The following tests will be done at each visit:
* A health assessment with a physical exam and review of life events and current health problems
* Blood, hair, and saliva samples
* Questionnaires about stress levels, personal health, and the caregiving process.
* Caregiver participants may have an optional fourth study visit within 72 hours after an ICU admission. This visit will include the same tests as the other visits....

DETAILED DESCRIPTION:
There are approximately 65.7 million unpaid caregivers in the United States with an estimated 8 percent providing care to someone with cancer. Although benefit-finding has been reported, providing care to a spouse or loved one with cancer is stressful and can have negative consequences for an individual s psychological and physical health. In cancer caregivers, studies have documented negative outcomes including symptoms of fatigue, impaired sleep quality, poor quality of life, anxiety and depression. These outcomes are of particular concern when cancer patients receive intense treatment such as hematopoietic stem cell transplantation (HSCT) where caregivers are embedded in a treatment trajectory that can extend 4 12 months. In dementia caregivers, additional outcomes have been reported including poor health habits and impaired immunity. In addition, longitudinal studies have also reported caregivers have an increased risk of morbidity and mortality, particularly from cardiovascular disease.

The stress response is initiated in the brain, which determines both the physiological and behavioral responses to an event. The normal physiologic response is complex and dynamic process by which the body responds to daily events in an effort to maintain equilibrium. If the stress becomes overwhelming for the individual, either due to the number or magnitude of stressors, the burden or overload can lead to dysregulation of biologic mediators and behavioral changes (poor sleep, eating or drinking too much, smoking, lack of physical activity) that can exacerbate disease (e.g. cardiovascular disease). A recent study in cancer caregivers demonstrated marked changes in neurohormonal and inflammatory processes in the year following a loved one s cancer diagnosis which may place the caregiver at risk for morbidity and mortality from disease. The relationships among the physiologic and psychological responses as well as behavioral changes to stress have not been explored in HSCT caregivers.

What is clear from the literature is that caregiving is stressful, and it appears to increase one s risk for morbidity and mortality, particularly by increasing cardiovascular risk. What is less clear is what behavioral, psychological, physiological and clinical changes are associated with the process of caregiver for individuals undergoing allogeneic HSCT, a particularly long and stressful experience. The purpose of this exploratory, pilot study is threefold: to longitudinally examine physiological, behavioral and clinical factors in HSCT caregivers during the acute transplant recovery period, to compare those factors in HSCT caregivers to non-caregivers, and to explore the associations among physiological, psychological, behavioral and clinical factors in HSCT caregivers.

Subjects will be accrued to this protocol if they are adult caregivers for a transplant recipient participating in their first allogeneic HSCT protocol at the Clinical Center. An equal sample of healthy volunteers that are non-caregivers will be recruited to serve as control subjects. A sample of 40 subjects (20 caregiver and 20 non-caregiver volunteers) will be recruited to capture the essence of the experience and adequately explore this population.

Each caregiver participant will have data collected prior to the recipient s HSCT (day 0), during the first week of outpatient visits following the recipient s initial discharge from the inpatient setting, and finally 6 weeks post the transplant recipients initial discharge from the hospital. Questionnaires will capture the psychological and behavioral outcomes and include: Caregiver Reaction Assessment (caregivers only), Health-Promoting Lifestyle Profile II, Perceived Stress Scale, The UCLA Loneliness Scale (Version 3), General Self-Efficacy Scale, and PROMIS Short Forms for Anxiety, Depression, Sleep disturbance and Fatigue. Clinical variables (e.g. vital signs) and physiological variables (e.g. cortisol) will be collected along with the questionnaires during the clinic visit and following history and physical exam by a Licensed Independent Practitioner (LIP). A sample of non-caregivers will be minimally matched for age, gender, and race/ethnicity, and complete all study procedures except the questionnaires that are specific to the caregiver s experience (e.g. caregiver burden). There will be no long term follow-up after the study participation period. Exploratory, hypothesis generating analyses will be performed using parametric and non-parametric techniques.

ELIGIBILITY:
* INCLUSION CRITERIA:

Caregiver Subjects

* Age greater than or equal to 18 years old
* Ability to comprehend the investigational nature of the study
* Able to read and speak English or Spanish
* Agrees to participate in the study
* Intends to serve as an active caregiver for a patient undergoing their 1st allogeneic HSCT at the NIH Clinical Center

Non-Caregiver Subjects

* Age greater than or equal to 18 years old
* Ability to comprehend the investigational nature of the study and provide informed consent
* Able to read and speak English or Spanish
* Agrees to participate in the study
* Match caregiver subject based on age, gender, and race/ethnicity.

If more than one caregiver is planned for the transplant recipient during the transplant phase, all caregivers will be invited to participate in the study. An active caregiver is defined as someone who lives with (at least 6 hours/day) the HSCT recipient during the study period (pre-HSCHT through 6 weeks post-discharge).

EXCLUSION CRITERIA: (all subjects)

* Age less than or equal to 18 years old
* Pregnant or lactating women
* Inability to comprehend investigational nature of study
* Inability to provide informed consent
* Unable to read and speak English or Spanish
* Does not agree to participate in study or follow study design (Beta)
* Glucocorticosteroid treatment in the last 2 months
* Diagnosis of Cushing, Addison or Parkinson s disease
* Prior heart transplant, have a pacemaker, diagnosis of orthostatic hypotension or autonomic dysfunction
* Smokers unwilling to cease smoking for at least 12 hours before specimen collection
* Unwilling to cease alcohol consumption for at least 24 hours before specimen collection
* Serving as a paid caregiver for any individual
* Serving as the HSCT donor (undergoing Stem Cell Mobilization)

EXCLUSION CRITERIA NON-CAREGIVER SUBJECTS:

Experienced a stressful life event in the preceding 3 months before enrollment (as determined by the following pre-screening questions:

In the last 3 months have you experienced?

* A serious illness, yourself or with someone close to you?
* Death of someone close?
* Faced imprisonment for yourself or someone close or had legal difficulties?
* Been unemployed or had a change in your work?
* Moved from your home or remodeled your home?
* Been involved in a natural disaster?
* A change in your marital status?
* A pregnancy, birth, miscarriage, or stillbirth?

Currently receiving mental health services or taking psychiatric medications

Currently or in the last 3 months served as a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09-26; Study Completion 2017-09-28

PRIMARY OUTCOMES:
To compare physiological factors and biomarkers of cardiovascular illness among HSCT caregivers during the acute transplant recovery period to non-caregivers. | 6 weeks

SECONDARY OUTCOMES:
To examine associations among physiological variables (salivary cortisol, norepinephrine, epinephrine, hs-CRP, TNF, and hs-IL6) and psychological health and healthy behaviors in HSCT caregivers. | 6 weeks
To characterize caregivers with no change and those with a change (in physiological or clinical factors) by demographic and HSCT recipient clinical factors. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Bevans, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hodges LJ, Humphris GM, Macfarlane G. A meta-analytic investigation of the relationship between the psychological distress of cancer patients and their carers. Soc Sci Med. 2005 Jan;60(1):1-12. doi: 10.1016/j.socscimed.2004.04.018. PMID 15482862
- [Background] Northouse LL, Katapodi MC, Song L, Zhang L, Mood DW. Interventions with family caregivers of cancer patients: meta-analysis of randomized trials. CA Cancer J Clin. 2010 Sep-Oct;60(5):317-39. doi: 10.3322/caac.20081. Epub 2010 Aug 13. PMID 20709946
- [Background] Burton LC, Newsom JT, Schulz R, Hirsch CH, German PS. Preventive health behaviors among spousal caregivers. Prev Med. 1997 Mar-Apr;26(2):162-9. doi: 10.1006/pmed.1996.0129. PMID 9085384